CLINICAL TRIAL: NCT04865471
Title: Resection And Partial Liver Segmental Transplantation With Delayed Total Hepatectomy as Treatment for Selected Patients With Unresectable Liver Metastases From Colorectal Carcinoma
Brief Title: Resection And Partial Liver Segmental Transplantation With Delayed Total Hepatectomy
Acronym: RAPID-Padova
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera di Padova (Other)
Collaborators: Istituto Oncologico Veneto IRCCS (Other)
Responsible Party: Principal Investigator, Prof. Umberto Cillo, Prof, Azienda Ospedaliera di Padova
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AOP1838
Record Dates: First submitted 2021-02-23; First posted 2021-04-29 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Liver Metastases
Keywords: Colorectal Liver Metastases; Auxiliary Liver Transplant
MeSH Terms: interventions — Liver Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Liver transplantation (Experimental): Auxiliary liver transplantation and staged hepatectomy
  Interventions: Procedure: Liver transplantation

INTERVENTIONS:
Procedure: Liver transplantation — Auxiliary liver transplantation and staged hepatectomy

SUMMARY:
RAPID is an auxiliary liver transplantation where a small liver partial graft (namely left lateral segments from living or cadaveric donors) is implanted orthotopically after a left hepatectomy of the native liver. Subsequently, in order to implement a fast regeneration of the transplanted segments a portal flow diversion is operated in the direction of the future remnant. After obtaining a fast regeneration of the auxiliary future remnant liver the native liver hepatectomy is completed as in a two stage- hepatectomy. Peculiar inclusion criteria will be adopted for patient selection with particular reference to the admission of patients with <3 lung metastases radically treated before transplantation.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 and <70 years
* Performance status, ECOG 0-1
* Histologically proved adenocarcinoma in colon or rectum
* BRAF wild-type CRC on primary tumor or liver metastases
* High standard oncological surgical resection of the primary tumor
* Liver metastases not eligible for curative liver resection confirmed by the validation committee
* At least one line (3 months) of chemotherapy
* At least 6 months time span from CRC resection and date of being listed on the transplantation list.
* At least 8 weeks of tumor control: stable disease or partial response according to RECIST 1.1 criteria
* No signs of extra hepatic metastatic disease or local recurrence on CT, MRI and Pet-CT except patients may have <3 lung lesions all<15mm resected or treated by radiotherapy or metastatic hilar nodes treated by resection and without recurrence at 3 months from resection or radiotherapy.
* Satisfactory blood tests creatinine in normal level, PLT >60.000/mm3, GB>2500/mm3
* CEA stable or in decrease
* Signed informed consent and expected cooperation of the patients for the treatment and follow up

Exclusion Criteria:

* Weight loss >10% the last 6 months
* Patient BMI > 30
* Participation refusal
* General contraindication to LT
* Other malignancies in the previous 5 years
* Pregnancy or breast feeding
* Any reason why, in the opinion of the investigator, the patient should not participate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Percent of transplanted patients receiving second stage hepatectomy within 4 weeks of segment 2/3 transplantation | within 4 weeks from liver transplantation
  Rate of second stage hepatectomy performed within 4 weeks from transplatation

SECONDARY OUTCOMES:
Intention to treat survival after liver transplantation | 3 and 5 years
  Time from transplantation to either death or censoring
Progression free survival | 3 and 5 years
  Time from enrolement to either progression or censoring
Proportion of drop out | within 100 days from listing
  Rate of drop out from listing
Mortality | within 90 days from second stage hepatectomy
  Rate of death within 90 days after second stage hepatectomy
Complication rate | within 90 days after liver transplant
  Complications according to Dindo Clavien Classification

CONTACTS AND LOCATIONS:
Locations (1):
- U.O.C Chirurgia Epatobiliare e Trapianti Epatici, Azienda Ospedaliera di Padova, Padua, Italy

IPD SHARING:
Plan to Share IPD: Undecided